CLINICAL TRIAL: NCT02173678
Title: A Randomized, Placebo-controlled, Double-blind, 3 Way Cross-over Safety and Tolerability Study of Single and Repetitive Dosing of COMBIVENT® HFA Compared to COMBIVENT® CFC and Placebo HFA in Healthy Male and Female Subjects (Cumulative Dose: 1600 mcg (HFA) or 1648 mcg (CFC) of Salbutamol Sulfate, 288 mcg of Ipratropium Bromide)
Brief Title: Safety and Tolerability of COMBIVENT® HFA as Compared to COMBIVENT® CFC and Placebo HFA in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1012.24
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-06

CONDITIONS: Healthy

ARMS (3):
- COMBIVENT® HFA (Experimental)
  Interventions: Drug: COMBIVENT® HFA-MDI
- COMBIVENT® CFC (Active Comparator)
  Interventions: Drug: COMBIVENT® CFC-MDI
- Placebo HFA-MDI (metered dose inhaler) (Placebo Comparator)
  Interventions: Drug: Placebo HFA-MDI

INTERVENTIONS:
Drug: COMBIVENT® HFA-MDI
  Arms: COMBIVENT® HFA
Drug: COMBIVENT® CFC-MDI
  Arms: COMBIVENT® CFC
Drug: Placebo HFA-MDI
  Arms: Placebo HFA-MDI (metered dose inhaler)

SUMMARY:
Study to assess the safety and tolerability of COMBIVENT® hydrofluoroalkane (HFA) as compared to COMBIVENT® chlorofluorocarbons (CFC) and placebo HFA after single and repetitive dosing in healthy male and female subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy males/females
* Age range from 21 to 50 years and be within 20% of their normal weight (Broca-Index)
* All female volunteers must use a safe contraception (i.e. oral contraceptives, intrauterine devices; sterilised) and must have a negative urine pregnancy test
* All subjects must have a negative hepatitis B, C and HIV tests as well as a negative drug screening
* Prior to admission to the treatment after giving his/her informed consent (in accordance with Good Clinical Practice and local legislation) in writing, each subject will have his/her medical history taken and will receive a complete medical examination (incl. blood pressure and pulse rate measurements) as well as 12-lead ECG within 14 days before the first administration of the test drug. Haematopoietic, hepatic and renal function tests will be carried out in the laboratory. The subject will fast for 12 hours before collection of specimens for all laboratory parameters
* Currently non-smoking (smoke free for >= one year and <=5 pack year smoking history)
* Normal spirometry as evidenced by a baseline FEV1 >= 90% of predicted normal value for age, height and sex
* Predicted normal values will be calculated according to European Community for Steel and Coal (ECCS)
* Ability to adequately use an inhalation aerosol device
* Ability to perform technically satisfactory pulmonary function tests

Exclusion Criteria:

* Volunteers will be excluded from the study if the results of the medical examination or laboratory test (especially serum glutamate oxaloacetate transaminase (SGOT) > 2-fold of upper normal range, serum glutamate pyruvate transaminase (SGPT) > 1.5 - fold of upper normal range) are judged by the investigator to differ significantly from normal clinical values
* Volunteers who have an eosinophil count >= 600/mm³. A repeat eosinophil count will not be conducted in these subjects
* Volunteers with a serum potassium value >+- 10% outside the normal range
* Volunteers with known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic immunological or hormonal disorders
* Volunteers with diseases of the central nervous system (such as epilepsy) or with psychiatric disorders
* Volunteers with known history of orthostatic hypotension, fainting spells or blackouts
* Volunteers with chronic or relevant acute infections
* Volunteers with upper respiratory tract infection in the past six weeks prior to the screening visit or between the screening visit and first test day
* Volunteers with a history of asthma or allergic rhinitis
* Volunteers with history of allergy/hypersensitivity (including drug allergy, especially anticholinergics and beta-agonist agents) which is deemed relevant to the trial as judged by the investigator
* Volunteers with known narrow-angle glaucoma
* Volunteers with disturbed micturition
* Volunteers who have taken a drug with a long half-life (>= 24 hours) within ten half-lives of the respective drug before enrolment in the study
* Volunteers who received any concomitant therapy, including over the counter medications (including vitamins, supplements and/or nonsteroidal antiinflammatory drugs; excluding oral or depository contraceptives) within one week of the screening visit
* Volunteers who have participated in another study with an investigational drug within the last two months preceding this study
* Volunteers who drink more than 40g of alcohol per day
* Volunteers who are dependent on drugs
* Volunteers who have donated blood (>= 100 ml ) within the last four weeks
* Volunteers who participated in excessive physical activities (e.g. competitive sports) within the last week before the study
* Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (i.e. contraceptives, intrauterine devices, sterilised)
* Volunteers with significant tremor measured on screening visit
* Previous participation in this study

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 1999-10; Primary Completion 1999-11 (Actual)

PRIMARY OUTCOMES:
Potential bronchoconstriction, objectively assessed by FEV1 and the occurence of cough, wheeze and shortness of breath | Baseline, 15, 50 , 85, 120, 155, 170, 200, 230, 260, 320 min. after first inhalation
Forced expiratory volume in one second (FEV1) | Baseline, 15, 50 , 85, 120, 155, 170, 200, 230, 260, 320 min. after first inhalation
Peak expiratory flow (PEF) | Baseline, 15, 50 , 85, 120, 155, 170, 200, 230, 260, 320 min. after first inhalation
Forced Vital Capacity (FVC) | Baseline, 15, 50 , 85, 120, 155, 170, 200, 230, 260, 320 min. after first inhalation
Mean maximal expiratory flow over the middle 50% of the FVC (MMEF25/75) | Baseline, 15, 50 , 85, 120, 155, 170, 200, 230, 260, 320 min. after first inhalation
Changes in serum potassium levels | Baseline, 85, 120, 155, 170 , 200, 230, 260 min after first inhalation
Occurence of adverse events | up to 30 days
Changes in blood pressure | Baseline, 15, 50 , 85, 120, 155, 170, 200, 230, 260, 320 min. after first inhalation
Changes in pulse rate | Baseline, 15, 50 , 85, 120, 155, 170, 200, 230, 260, 320 min. after first inhalation
Changes in respiratory rate | Baseline, 15, 50 , 85, 120, 155, 170, 200, 230, 260, 320 min. after first inhalation
Tremor measurement | Baseline, 15, 50 , 85, 120, 155, 170, 200, 230, 260, 320 min. after first inhalation
Changes in electrocardiogram (ECG), QTc interval | Baseline, 85, 120, 155, 170, 200 min after first inhalation (230, 260, 320 min only to be performed if abnormal ECG)
Number of subjects with clinically relevant changes from baseline in physical examination | Screening, end-of study-evaluation (within 8 days after the last treatment)
Number of subjects with clinically signification changes from baseline in laboratory values | Screening, end-of study-evaluation (within 8 days after the last treatment)